CLINICAL TRIAL: NCT05939401
Title: ANCABio - a Study Regarding Tumour Microenvironment and the Predictive Capability of Biopsies from Anal Cancer in Predicting Response and Outcome
Brief Title: A Study Regarding Tissue Response During and After Treatment for Anal Cancer
Acronym: ANCABio
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Other Study IDs: ANCABio
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Anal Cancer
Keywords: Anal cancer, Tumour micro environment, Chemoradiotherapy
MeSH Terms: conditions — Anus Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumour tissue, adjacent normal tissue, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Biopsies — Biopsies and blood samples will be taken at time of diagnosis or recurrence

SUMMARY:
The aim of this study is to improve the understanding for the tumour biology in relation to treatment response in patients with anal cancer by examining:

* The tumour microenvironment
* The localisation of and cellular interactions between the tumour and immune cells
* The gene and protein expression by cells present in the tumour and surrounding tissue.

DETAILED DESCRIPTION:
All adult patients with anal cancer presenting within the Sahlgrenska University Hospital catchment area or treated at any time at Sahlgrenska University Hospital are eligible and will be asked to participate. The patients that are newly diagnosed or that have a suspected recurrence will be offered to enter the study with biopsies as well as blood samples during the diagnostic examination that is performed under anaesthesia. Biopsies will then be taken during follow-up exams if applicable. Biopsies will also be taken during surgery if that is scheduled and in cases where surgery is not necessary biopsies will be taken if the patient undergoes examinations under anaesthesia after treatment cessation.

If it is not possible to take biopsies prior treatment blood samples will still be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent anal cancer

Exclusion Criteria:

* No diagnosis of anal cancer, contraindication to biopsies and blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to Sahlgrenska University Hospital with anal cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Tumour micro environment | 2024-2029
  Evaluation of immuncell infiltrates in the tumour micro environment
ctDNA | 2024-2029
  circulating tumour DNA

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg
  - Sahlgrenska University Hospital, Gothenburg

IPD SHARING:
Plan to Share IPD: No